CLINICAL TRIAL: NCT07230730
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of SHR-1918 in Patients With Hyperlipidemia
Brief Title: A Trial to Evaluate the Efficacy and Safety of SHR-1918 in Patients With Hyperlipidemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1918-302
Record Dates: First submitted 2025-09-22; First posted 2025-11-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SHR-1918 low dose (Experimental)
  Interventions: Drug: SHR-1918
- SHR-1918 placebo low dose (Placebo Comparator)
  Interventions: Drug: SHR-1918 placebo
- SHR-1918 high dose (Experimental)
  Interventions: Drug: SHR-1918
- SHR-1918 placebo high dose (Placebo Comparator)
  Interventions: Drug: SHR-1918 placebo

INTERVENTIONS:
Drug: SHR-1918 — SHR-1918
  Arms: SHR-1918 high dose; SHR-1918 low dose
Drug: SHR-1918 placebo — SHR-1918 placebo
  Arms: SHR-1918 placebo high dose; SHR-1918 placebo low dose

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of SHR-1918 in reducing serum low-density lipoprotein cholesterol (LDL-C) and total triglycerides (TG) in patients with hyperlipidemia compared with placebo, and also includes To evaluate the effectiveness of SHR-1918 in reducing other lipid indicators in patients with mixed hyperlipidemia and to assess the safety of SHR-1918 in patients with mixed hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. the age must be at least 18 years old, and both men and women are eligible;
2. the patient was receiving a stable dose of statins at the time of screening,, and the fasting LDL-C met: For individuals with extremely high risk of ASCVD, LDL-C≥1.4 mmol/L; for those with very high risk of ASCVD, LDL-C≥1.8 mmol/L; and for those with medium and high risk of ASCVD, ≥2.6 mol/L;
3. Fasting TG≥2.3，and ≤5.6 mmol/L;
4. Understand the research procedures and methods, voluntarily participate in this trial and sign the informed consent form in person；

Exclusion Criteria:

1. poorly controlled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg) at the time of screening or before randomization；
2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or γ -glutamyl transferase (GGT) > 3× upper limit of normal (ULN), or total bilirubin > 2×ULN；
3. Thyroid stimulating hormone (TSH) is lower than the lower limit of normal (LLN) or greater than 1.5×ULN；
4. The estimated glomerular filtration rate (eGFR) is less than 30 mL/min/1.73m2；
5. Previously suffering from diseases that have a significant impact on blood lipid levels, such as nephrotic syndrome, severe liver diseases, Cushing's syndrome, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The percentage change of serum LDL-C from baseline; | Baseline and Week 24
The percentage change in serum TG from baseline; | Baseline and Week 24

SECONDARY OUTCOMES:
Percentage change of serum non-high-density lipoprotein cholesterol (non-HDL-C) from baseline; | Baseline and Week 24
The percentage change in serum total cholesterol (TC) from baseline; | Baseline and Week 24
The percentage change of serum apolipoprotein B (ApoB) from baseline at week 24; | Baseline and Week 24
The percentage change of serum apolipoprotein A1 (ApoA1) from baseline; | Baseline and Week 24
The change from baseline in serum LDL-C； | Baseline and Week 24
The change from baseline in serum TG； | Baseline and Week 24
The change from baseline in serum non-HDL-C； | Baseline and Week 24
The change from baseline in serum TC； | Baseline and Week 24
The change from baseline in serum ApoB； | Baseline and Week 24
The change from baseline in serum ApoA1； | Baseline and Week 24
Absolute and relative percent change from baseline in serum lipoprotein(a) (Lp(a)); | Baseline and Week 24
Absolute and relative percent change from baseline in serum high-density lipoprotein cholesterol (HDL-C); | Baseline and Week 24
LDL-C goal attainment rates at Week 24, overall and by risk subgroup; | Baseline and Week 24
Absolute and percentage change from baseline in serum non-HDL-C at Week 48; | Baseline and Week 48
Absolute and percentage change from baseline in serum ApoB at Week 48; | Baseline and Week 48
Absolute and percentage change from baseline in serum Lp(a) at Week 48; | Baseline and Week 48
Absolute and percentage change from baseline in serum TC at Week 48; | Baseline and Week 48
Absolute and percentage change from baseline in serum TG at Week 48; | Baseline and Week 48
Absolute and percentage change from baseline in serum HDL-C at Week 48; | Baseline and Week 48
Absolute and percentage change from baseline in serum ApoA1 at Week 48; | Baseline and Week 48
LDL-C goal attainment rates at Week 48, overall and by risk subgroup | Baseline and Week 48
The incidence and severity of adverse events (AEs) throughout the study; | up to week 52
Injection site reactions (pain, pruritus, erythema, swelling, induration, and rash) throughout the study; | up to week 52
Major adverse cardiovascular events (Cardiovascular death, Non-fatal myocardial infarction, Non-fatal stroke and Coronary revascularization) throughout the study; | up to week 52

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided